CLINICAL TRIAL: NCT00330655
Title: An Open-Label, Prospective Trial of Memantine in the Treatment of Moderate to Severe Binge Eating Disorder Associated With Obesity
Brief Title: An Open-Label Trial of Memantine in the Treatment of Binge Eating Disorder
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Mclean Hospital (Other)
Collaborators: Forest Laboratories (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2006-P-000296/1
Record Dates: First submitted 2006-05-25; First posted 2006-05-29 (Estimated); Last update posted 2007-08-14 (Estimated); Status verified 2007-08

CONDITIONS: Binge Eating Disorder
Keywords: Binge eating; Obesity; Eating disorder
MeSH Terms: conditions — Binge-Eating Disorder; Bulimia; Obesity; Feeding and Eating Disorders | interventions — Memantine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: memantine

SUMMARY:
We hypothesize that memantine may be a safe and effective treatment for moderate to severe binge eating disorder associated with obesity.

During this 12-week, open-label, outpatient study, male and female subjects between the ages of 18 and 65 years who have moderate to severe binge eating disorder and are obese will be treated with open-label memantine. Following this 12-week treatment phase, subjects may be eligible to continue into an extension phase which will last an additional 12 weeks. During the extension phase subjects will continue open-label memantine treatment.

DETAILED DESCRIPTION:
Binge eating disorder is a newly recognized disorder characterized by recurrent episodes of binge eating without extreme behaviors to lose weight characteristic of bulimia nervosa or anorexia nervosa and it is associated with overweight and obesity in both clinical and community populations. Preliminary clinical data from a recent, small, 5-week, open-label therapeutic trial in obese patients with binge eating disorder in Germany found memantine to be effective in weight reduction and reduction of binge episodes.

We plan to study 15 male and female subjects between the ages of 18 and 65 years who have binge eating disorder (with 3 or more binge days per week in the 2 weeks prior to baseline) and have a body mass index (BMI) between 30 and 50 kg/m2. During the 12-week treatment phase subjects will receive open-label memantine titrated up to 20mg/day, or the subjects maximum tolerated dose. Upon completion of the treatment phase, subjects will either taper their study medication and return for a final post-taper visit or continue on their current dose of study medication in the 12-week extension phase.

ELIGIBILITY:
Inclusion Criteria:

* Subjects may be male or female, 18-65 years old
* Diagnosis of binge eating disorder
* Subjects must have 3 or more binge days per week for the two weeks prior to the start of the study
* Subjects must have a BMI between 30 and 50 kg/m2

Exclusion Criteria:

* Current or lifetime history of schizophrenia, other psychotic disorder, or bipolar disorder
* Subjects with a history of a personality disorder
* Subjects with clinically significant depression
* Subjects with substance use of dependence
* Subjects who are pregnant or lactating
* Subjects with a serious medical condition

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2006-05; Study Completion 2007-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James I Hudson, M.D., Sc.D., Principal Investigator — Mclean Hospital
Locations (1):
- McLean Hospital, Belmont, Massachusetts, United States